CLINICAL TRIAL: NCT00841516
Title: A Multicentre Randomised Placebo-controlled Double-blind Clinical Trial for the Immunological and Histological Evaluation of Specific Immunotherapy With an Aluminium Hydroxide-adsorbed Recombinant Hypoallergenic Derivative of the Major Birch Pollen Allergen, rBet v1-FV
Brief Title: Immunological and Histological Evaluation of Specific Immunotherapy With Recombinant Hypoallergenic Derivative
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AL0801rB; 2008-006258-16 (EudraCT Number)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Specific immunotherapy; SIT; SCIT; recombinant; Type 1 - Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo was given the same way as a subcutaneous (just under the skin) injection.
  Interventions: Other: Placebo
- 80 µg rBet v1-FV Immunotherapy (Experimental): All randomized patients were treated with either placebo or 80 µg rBet v1-FV (maintenance dose) for 2 years.
  Interventions: Biological: rBet v1-FV

INTERVENTIONS:
Other: Placebo — Placebo was given the same way as a subcutaneous (just under the skin) injection.
  Other Names: Comparator
  Arms: Placebo
Biological: rBet v1-FV — Placebo was given the same way as a subcutaneous (just under the skin) injection.
  Other Names: Specific Immunotherapy
  Arms: 80 µg rBet v1-FV Immunotherapy

SUMMARY:
This trial is performed for the immunological and histological evaluation of specific immunotherapy with an aluminium hydroxide-adsorbed recombinant hypoallergenic derivative of the major birch pollen allergen, rBet v1-FV

DETAILED DESCRIPTION:
Type I allergy is an immune-disorder which stems from the formation of IgE antibodies against proteins and glycoproteins from plants, insects, animals and fungi, most of which are normally considered harmless. The cross-linking of specific IgE antibodies on effector cells by allergens activates an immunological cascade leading to the symptoms of Type I allergy including rhinitis, conjunctivitis, asthma, and anaphylactic shock. Allergic Rhinitis is the most common chronic atopic disease and is associated with considerable cost and co-morbidity. Seasonal allergic rhinitis (SAR), triggered by pollen from trees, grasses and weeds, is characterized by sneezing, nasal congestion, nasal itching, rhinorrhea, and pruritic, watery, red eyes.

Recombinant preparations offer various advantages over those based on natural allergen extracts. Recombinant proteins can be produced in highly purified forms of pharmaceutical quality; proteins are molecularly defined thus ensuring product consistency and minimising problems related to allergen extract standardisation; preparations only include those proteins that are considered relevant for specific immunotherapy; the risk of contamination with other allergenic material is excluded; the whole production process can be designed to exclude any risk factors for the introduction of infectious agents; the relative dosages of individual components of a final preparation can be optimised to favour better clinical efficacy. Allergy vaccination (AV) mediates the immune response to allergen exposure by altering the TH2 response in favour of a TH1 T-cell response, increasing IgG production and decreasing the production of inflammatory cytokines. rBet v1-FV is an AV designed to enhance beneficial immune responses. The investigational product has demonstrated efficacy and good tolerability in one previous pivotal Phase III and two previous Phase II studies.

ELIGIBILITY:
Inclusion Criteria:

* Positive SPT
* Positive EAST
* Positive specific provocation test

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Changes in populations of inflammatory cells and subpopulations of immunologically active cells. | Cells were obtained before and after one year of treatment with rBet v1-FV.
  All these cells were evaluated in nasal biopsies obtained before the start of treatment (outside the birch pollen season) and during immunotherapy (after one year of treatment with rBet v1-FV) around the peak of the pollen season.

SECONDARY OUTCOMES:
Immunologic changes | 4 time points.
  Specific IgE, IgG1 and IgG4 were measured at 4 points: at screening visit (V I/1), after uptitration (V II/10) and after birch pollen season in first and second treatment year (V II).

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Rak, Prof.Dr.med., Principal Investigator — Prof. Dr. med. Rak
Locations (1):
- Prof. Dr. med. Sabina Rak, Gothenburg, Sweden

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-006258-16/SE